CLINICAL TRIAL: NCT04860180
Title: Effect of Surgical or Conservative Approach in Patients With Adrenal Incidentalomas on Cardiovascular, Metabolic, Neuropsychological and Bone Manifestations: Respective Roles of Cortisol Secretion and Glucocorticoid Sensitivity
Brief Title: Effect of Surgical or Conservative Approach in Patients With Adrenal Incidentalomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Casa Sollievo della Sofferenza IRCCS (Other); I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other); Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Iacopo Chiodini, Associate Professor of Endocrinology, MD, Istituto Auxologico Italiano
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RF-2013-02356606
Record Dates: First submitted 2021-02-16; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Adrenal Incidentaloma; Subclinical Hypercortisolism
MeSH Terms: conditions — Adrenal incidentaloma | interventions — Adrenalectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A, surgery (Experimental): adrenalectomy
  Interventions: Procedure: adrenalectomy
- B, observation (No Intervention): conservative follow up

INTERVENTIONS:
Procedure: adrenalectomy
  Arms: A, surgery

SUMMARY:
Subclinical hypercortisolism (SH) is a status of asymptomatic hypercortisolism, frequently found in patients with adrenal adenomas (estimated prevalence: 0.8-2% after 60 years of age). Although SH may lead to diabetes, hypertension and osteoporosis, the diagnostic SH criteria and those suggesting the need of adrenalectomy are debated. Indeed, beside the cortisol secretion, the individual cortisol sensitivity may play a role in determining the SH consequences.

Subjects with possible SH due to adrenal adenoma will be randomized to surgery/conservative follow up. The effects of surgery on the cardiovascular, bone, metabolic complications of SH and on neuropsychological aspects and quality of life (QoL) and the possibility to predict them by using cortisol sensitivity and secretion markers will be studied. The study may clarify how to individuate patients who can benefit from surgery. These results will help reducing the costs of both useless surgical operations and SH consequences.

DETAILED DESCRIPTION:
Subclinical hypercortisolism (SH) is a status of asymptomatic hypercortisolism, which is present in up to the 30% of patients with incidentally discovered adrenal adenomas (adrenal incidentalomas, AI). Since AI are present in 7-10% of individuals after 60 years of age, the estimated SH prevalence in this population is 0.8-2%. In patients with SH due to an adrenal adenoma the risk of diabetes, hypertension, cardiovascular events, osteoporosis and mortality seems to be increased, and monolateral adrenalectomy beneficial. However, no randomized studies evaluated the effects of surgery on SH consequences and established the criteria indicating the need of surgery itself. Thus, in many patients the SH diagnosis is uncertain and the best approach (surgical or conservative) unknown. These uncertainties are also due to the influence of the individual glucocorticoid (GC) sensitivity. Indeed, in the single individual the various polymorphisms of GC receptor (GR) and the different 11ß-hydroxysteroid-dehydrogenase type 2 enzyme (11HSD2) activity, regulating the tissue exposure to the active GC, may differently predispose to the consequences of GC excess. Therefore, in AI patients, beside the evaluation of the degree of the cortisol hypersecretion, the assessment of the cortisol sensitivity may be useful in establishing the individual risk of SH consequences and the possible usefulness of a surgical approach.

Specific Aim:

In AI subjects with uncertain SH the combined evaluation of the clinical features together with the parameters of cortisol secretion and sensitivity will consent to decide which patient has the greatest probability to ameliorate after surgery.

1. To assess the variation of blood pressure control, lipids and glucose metabolism, vascular damage, bone mineral density (BMD), clinical and morphometric vertebral fractures, body composition, coagulation parameters, neuropsychological aspects and quality of life (QoL) in AI patients with uncertain SH after the surgical removal of the adrenal mass or after a conservative treatment.
2. To assess in AI patients and uncertain hypercortisolism the effect of the surgical and conservative approach on cardiovascular, metabolic and bone manifestations, neuropsychological aspects and quality of life (QoL), in relation to the degree of cortisol secretion and sensitivity.
3. To establish the best clinical-biochemical criteria for diagnosing SH, on the basis of the changes of the outcomes after the surgical or conservative approach, and therefore, for addressing the treatment of choice in the individual patient with AI.

Methods. During the enrollment period (24 months), all patients between 40 and 75 years of age referred for unilateral AI larger than 1 cm will be evaluated.

In all subjects, adrenocorticotroph hormone (ACTH), urinary free cortisol (UFC), cortisol after 1-mg overnight dexamethasone suppression test (1mgDST) and the GR polymorphisms of N363S, BclI and ER22/23EK will be assessed. Patients with 1mgDST >1.8 mcg/dL will undergo a low dose (2 mg for 2 days) dexamethasone suppression test (LDDST). Patients with 1mgDST and LDDST >5 mcg/dL and suppressed (<5 pg/mL) ACTH levels will be excluded as affected by biochemically overt hypercortisolism, that requires surgery. AI patients with 1mgDST or LDDST <1.8 mcg/dL will be excluded as certainly not affected with SH. AI patients with AI >5 cm will leave the study as in this case surgery is mandatory.

Eventually, after the enrollment period, 54 AI patients with uncertain SH will be included and randomized to surgery (Group1) or conservative treatment (Group 2). The follow-up period will last 24 months (after withdrawal of GC substitution therapy, if needed, for Group 1). Group 1 patients will undergo laparoscopic or laparotomic adrenalectomy, depending on the AI size and their clinical characteristics.

Evaluations at baseline, 6, 12 and 24 months: blood pressure (BP), body weight (BW), body mass index (BMI), waist circumference, glucose, lipid and coagulation parameters, body composition and adenoma size by CT (Group 2 patients).

Group 2 patients with a >1 cm adenoma increase or appearance of overt SH will leave the study. At baseline and after 24 months, bone mineral density (BMD) and quality (by trabecular bone score, TBS), vertebral fractures (VFx), carotid atherosclerosis, neuropsychological aspects and QoL, will be assessed.

The patients will be defined: i) obese, in the presence of BMI >30 kg/m2; ii) hypertensive in the presence of systolic BP >130 mmHg and/or diastolic BP >85 mmHg and/or any antihypertensive treatment; iii) diabetic, in the presence of the World Health Organization criteria, and/or any hypoglycemic drug, iv) dyslipidemic, in the presence of triglyceride levels >150 mg/dl or high-density lipoprotein (HDL) cholesterol levels <40 or 50 mg/dl in males and females, respectively.

The improvement/worsening during follow-up will be defined as follows: for obesity in the presence of a >5% BW decrease/increase, for hypertension if the non-hypertensive patients passed from a pre-hypertension category to another or the hypertensive patients from a hypertension grade to another; for diabetes and dyslipidemia if fasting glucose and cholesterol levels pass from a category to another, respectively, following the Adult Treatment Panel III criteria.

The efficacy of the surgical and conservative approach on the basis of the changes of BP, BW, glucose and lipid control, BMD, VFx incidence (primary outcomes) will be compared. The effect of surgery on the coagulation parameters, carotid atherosclerosis, body composition, neuropsychological aspects and QoL (secondary outcomes) will be also evaluated.

At baseline, and at 6, 12 and 24 months, beside ACTH, 1mgDST and UFC, the midnight salivary cortisol (MSalC) and urinary free cortisone (UFCo) levels and the UFC/UFCo ratio (index of 11HSD2 activity) will be assessed In Group 1 and Group 2 patients the association between the changes of the primary and secondary outcomes with the cortisol secretion parameters and the presence/absence of GC sensitizing GR polymorphisms and the degree of 11HSD2 activity, will be evaluated.

An algorithm for predicting the effect of the surgical or conservative approach on the primary outcomes in the individual AI patient with uncertain SH. The algorithm, based on the combination of the SH complications at baseline (hypertension, osteoporotic fractures, diabetes) with the presence/absence of GC sensitizing GR polymorphisms, degree of 11HSD2 activity and parameters of cortisol secretion, will be retrospectively tested on the study population, will be elaborated. This would consent to evaluate positive and negative predictive value of the algorithm for predicting the response to surgery in the individual patient with AI.

ELIGIBILITY:
Inclusion Criteria:

* unilateral adrenal incidentaloma larger than 1 cm
* cortisol after 1-mg overnight dexamethasone suppression test (1mgDST) between 1.8 and 5 mcg/dl

Exclusion Criteria:

* hypogonadism, thyrotoxicosis, chronic renal failure and hepatic disease, alcoholism, eating, rheumatologic or hematological disorders;
* intake of drugs influencing cortisol and dexamethasone metabolism or cortisol secretion;
* signs of hypercortisolism (moon facies, striae rubrae, easy bruising);
* possible metastatic disease or radiologic features not consistent with adrenocortical adenoma at computed tomography (CT);
* pheochromocytoma and aldosteronoma;
* non-adrenal SH.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2016-09-29 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2022-12-08 (Estimated)

PRIMARY OUTCOMES:
variation of blood pressure | 6 months
  To assess the variation of blood pressure ambulatory systolic and diastolic blood pressure (BP, mmHg), and antihypertensive treatment at baseline and follow-up will be assessed; BP will be considered improved or worsened if the non-hypertensive patients passed from a pre-hypertension category to another or the hypertensive patients from a hypertension grade to another in accordance to giudelines, of if if antihypertensive treatment was reduced by 50%
variation of glucose levels | 6 months
  To assess the variation of glucose levels, fasting glucose levels and glucose levels after oral glucose tolerance test will be evaluated at baseline and follow-up. Glucose levels will be considered improved or worsened if fasting glucose levels pass from a category to another, following the Adult Treatment Panel III criteria or if antidiabetic treatment was reduced by 50%
variation of lipids | 6 months
  At baseline and follow up triglyceride levels; total cholesterol levels, HDL and LDL levels (mg/dl) will be evaluated. Dyslipidemia will be diagnosed in the presence of triglyceride levels >150 mg/dl or high-density lipoprotein (HDL) cholesterol levels <40 or 50 mg/dl in males and females. dyslipidemia will be defined improved or worsened if cholesterol levels pass from a category to another, following the Adult Treatment Panel III criteria
variation of body weight | 6 months
  At baseline and follow up body weight (kilograms) will be evaluated. the improvement/worsening during follow-up will be defined in the presence of a >5% BW decrease/increase
variation of bone mineral density (BMD) | 24 months
  To assess the variation of bone mineral density at baseline and follow-up a Dual-energy X-ray absorptiometry (DXA) scan will be performed
occurrence of vertebral fractures | 24 months
  A dorso-lumbar spine x-ray to evaluate the presence of morphometric fractures (presence/absence) will be performed
variation of intimal medial thickness | 12 months
  To assess the variation of vascular damage a supra-aortic trunk echo-Doppler to evaluate at baseline and follow-up variations of intimal medial thickness will be performed
variation of Relative wall thickness (RWT) | 12 months
  the variation of Relative wall thickness (RWT) will be evaluated by an echocardiography. It will be calculated from Left ventricular end diastolic dimension (LVEDD) (mm); Interventricular septal end diastole (IV Sd, mm) and Posterior wall thickness at end-diastole (PWd) parameters (mm)
variation of Sheehan Disability Scale | 6 months
  Sheehan Disability Scale will be evaluated to assess perceived stress (SDS-stress scale ranges 1-10, a higher score means higher levels of stress)
Cognitive evaluation by Brief Assessment Cognition in Schizophrenia (BACS) score | 6 months
  BACS evaluate verbal memory score (normal if >33); working memory (normal if >14.9); verbal fluency (normal if >31.6), symbol coding (normal if >40.5), tower of london (>12.4)

SECONDARY OUTCOMES:
cortisol secretion and sensitivity | 24 months
  To correlate the effect of the surgical and conservative approach in relation to the degree of cortisol secretion and sensitivity we will evaluate the GR polymorphisms of N363S, BclI and ER22/23EK ,midnight salivary cortisol (MSalC) and urinary free cortisone (UFCo) levels and the UFC/UFCo ratio (index of 11HSD2 activity)
variation of Inflammation markers and bone metabolism markers | 6 months
  irisine, Tumor Necrosing Factor (TNF)- alpha, interleukin (IL)-6, adiponectin, resistin, sclerostin, Dickkopf-related protein (DKK) 1, N-terminal propeptide of type 1 collagen (P1NP) , monocytechemoattractant protein 1 (CCL2/MCP-1) levels will be assessed (pg/ml). Paired samples T-test will be used to compare baseline and follow-up levels.

CONTACTS AND LOCATIONS:
Overall Officials: Iacopo Chiodini, Professor, Principal Investigator — Istituto Auxologico Italiano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reincke M. Subclinical Cushing's syndrome. Endocrinol Metab Clin North Am. 2000 Mar;29(1):43-56. doi: 10.1016/s0889-8529(05)70115-8. PMID 10732263
- [Background] Terzolo M, Bovio S, Reimondo G, Pia A, Osella G, Borretta G, Angeli A. Subclinical Cushing's syndrome in adrenal incidentalomas. Endocrinol Metab Clin North Am. 2005 Jun;34(2):423-39, x. doi: 10.1016/j.ecl.2005.01.008. PMID 15850851
- [Background] Chiodini I, Morelli V, Masserini B, Salcuni AS, Eller-Vainicher C, Viti R, Coletti F, Guglielmi G, Battista C, Carnevale V, Iorio L, Beck-Peccoz P, Arosio M, Ambrosi B, Scillitani A. Bone mineral density, prevalence of vertebral fractures, and bone quality in patients with adrenal incidentalomas with and without subclinical hypercortisolism: an Italian multicenter study. J Clin Endocrinol Metab. 2009 Sep;94(9):3207-14. doi: 10.1210/jc.2009-0468. Epub 2009 Jun 23. PMID 19549741
- [Background] Morelli V, Reimondo G, Giordano R, Della Casa S, Policola C, Palmieri S, Salcuni AS, Dolci A, Mendola M, Arosio M, Ambrosi B, Scillitani A, Ghigo E, Beck-Peccoz P, Terzolo M, Chiodini I. Long-term follow-up in adrenal incidentalomas: an Italian multicenter study. J Clin Endocrinol Metab. 2014 Mar;99(3):827-34. doi: 10.1210/jc.2013-3527. Epub 2014 Jan 1. PMID 24423350
- [Background] Di Dalmazi G, Vicennati V, Garelli S, Casadio E, Rinaldi E, Giampalma E, Mosconi C, Golfieri R, Paccapelo A, Pagotto U, Pasquali R. Cardiovascular events and mortality in patients with adrenal incidentalomas that are either non-secreting or associated with intermediate phenotype or subclinical Cushing's syndrome: a 15-year retrospective study. Lancet Diabetes Endocrinol. 2014 May;2(5):396-405. doi: 10.1016/S2213-8587(13)70211-0. Epub 2014 Jan 29. PMID 24795253
- [Background] Manenschijn L, van den Akker EL, Lamberts SW, van Rossum EF. Clinical features associated with glucocorticoid receptor polymorphisms. An overview. Ann N Y Acad Sci. 2009 Oct;1179:179-98. doi: 10.1111/j.1749-6632.2009.05013.x. PMID 19906240
- [Background] Szappanos A, Patocs A, Toke J, Boyle B, Sereg M, Majnik J, Borgulya G, Varga I, Liko I, Racz K, Toth M. BclI polymorphism of the glucocorticoid receptor gene is associated with decreased bone mineral density in patients with endogenous hypercortisolism. Clin Endocrinol (Oxf). 2009 Nov;71(5):636-43. doi: 10.1111/j.1365-2265.2009.03528.x. Epub 2009 Jan 22. PMID 19207316
- [Background] Tomlinson JW, Walker EA, Bujalska IJ, Draper N, Lavery GG, Cooper MS, Hewison M, Stewart PM. 11beta-hydroxysteroid dehydrogenase type 1: a tissue-specific regulator of glucocorticoid response. Endocr Rev. 2004 Oct;25(5):831-66. doi: 10.1210/er.2003-0031. PMID 15466942
- [Background] Eller-Vainicher C, Morelli V, Ulivieri FM, Palmieri S, Zhukouskaya VV, Cairoli E, Pino R, Naccarato A, Scillitani A, Beck-Peccoz P, Chiodini I. Bone quality, as measured by trabecular bone score in patients with adrenal incidentalomas with and without subclinical hypercortisolism. J Bone Miner Res. 2012 Oct;27(10):2223-30. doi: 10.1002/jbmr.1648. PMID 22549969
- [Background] Webb SM, Badia X, Barahona MJ, Colao A, Strasburger CJ, Tabarin A, van Aken MO, Pivonello R, Stalla G, Lamberts SW, Glusman JE. Evaluation of health-related quality of life in patients with Cushing's syndrome with a new questionnaire. Eur J Endocrinol. 2008 May;158(5):623-30. doi: 10.1530/EJE-07-0762. PMID 18426820
- [Background] Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Report of the expert committee on the diagnosis and classification of diabetes mellitus. Diabetes Care. 2003 Jan;26 Suppl 1:S5-20. doi: 10.2337/diacare.26.2007.s5. No abstract available. PMID 12502614
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Vidal J. Updated review on the benefits of weight loss. Int J Obes Relat Metab Disord. 2002 Dec;26 Suppl 4:S25-8. doi: 10.1038/sj.ijo.0802215. PMID 12457296
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Erdine S, Kiowski W, Agabiti-Rosei E, Ambrosioni E, Lindholm LH, Viigimaa M, Adamopoulos S, Agabiti-Rosei E, Ambrosioni E, Bertomeu V, Clement D, Erdine S, Farsang C, Gaita D, Lip G, Mallion JM, Manolis AJ, Nilsson PM, O'Brien E, Ponikowski P, Redon J, Ruschitzka F, Tamargo J, van Zwieten P, Waeber B, Williams B; Management of Arterial Hypertension of the European Society of Hypertension; European Society of Cardiology. 2007 Guidelines for the Management of Arterial Hypertension: The Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2007 Jun;25(6):1105-87. doi: 10.1097/HJH.0b013e3281fc975a. No abstract available. PMID 17563527
- [Background] Athimulam S, Delivanis D, Thomas M, Young WF, Khosla S, Drake MT, Bancos I. The Impact of Mild Autonomous Cortisol Secretion on Bone Turnover Markers. J Clin Endocrinol Metab. 2020 May 1;105(5):1469-77. doi: 10.1210/clinem/dgaa120. PMID 32154561
- [Background] Bancos I, Alahdab F, Crowley RK, Chortis V, Delivanis DA, Erickson D, Natt N, Terzolo M, Arlt W, Young WF Jr, Murad MH. THERAPY OF ENDOCRINE DISEASE: Improvement of cardiovascular risk factors after adrenalectomy in patients with adrenal tumors and subclinical Cushing's syndrome: a systematic review and meta-analysis. Eur J Endocrinol. 2016 Dec;175(6):R283-R295. doi: 10.1530/EJE-16-0465. Epub 2016 Jul 22. PMID 27450696
- [Derived] Morelli V, Frigerio S, Aresta C, Passeri E, Pugliese F, Copetti M, Barbieri AM, Fustinoni S, Polledri E, Corbetta S, Arosio M, Scillitani A, Chiodini I. Adrenalectomy Improves Blood Pressure and Metabolic Control in Patients With Possible Autonomous Cortisol Secretion: Results of a RCT. Front Endocrinol (Lausanne). 2022 Jun 2;13:898084. doi: 10.3389/fendo.2022.898084. eCollection 2022. PMID 35721734